CLINICAL TRIAL: NCT06477679
Title: Velopharyngeal Insufficiency Evaluation Post Cleft Palate Repair. Furlow With Buccinator Myomucosal Flap Versus Two Flap Palatoplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ragab Ahmed Ali, ASSISTANT LECTURE-pediatricSURGERY department-sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: soh-Med-24-05-02MD
Record Dates: First submitted 2024-06-10; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Cleft Palate
MeSH Terms: conditions — Cleft Palate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): . Furlow with buccinators myomucosal flap. Two opposing Z-plasties were designed on the oral and nasal mucosal surface. The posterior based flap on each surface was composed of muscle and mucosa, and the anterior surface was composed of mucosa only. BMFs were raised from the donor site, and immediately transferred to the recipient site to repair the defect. The flaps were sutured to the recipient site. The donor site was also closed primarily
  Interventions: Procedure: • Furlow with buccinators myomucosal flap
- group B (Active Comparator): • Two flap palatoplasty as von langenbeck technique, Upper left: Medial incisions design. Upper right: Lateral relaxing incisions and nasal mucosa closure using the anterior triangular flap and lateral nasal mucosa flaps. Release of the abnormal muscular insertion is performed. But two flap palatoplasty can lengthen the soft palate by push-back.
  Interventions: Procedure: • Two flap palatoplasty as von langenbeck technique

INTERVENTIONS:
Procedure: • Furlow with buccinators myomucosal flap — • Furlow with buccinators myomucosal flap. Two opposing Z-plasties were designed on the oral and nasal mucosal surface. The posterior based flap on each surface was composed of muscle and mucosa, and the anterior surface was composed of mucosa only. BMFs were raised from the donor site, and immediately transferred to the recipient site to repair the defect. The flaps were sutured to the recipient site. The donor site was also closed primarily
  Arms: group A
Procedure: • Two flap palatoplasty as von langenbeck technique — • Two flap palatoplasty as von langenbeck technique, Upper left: Medial incisions design. Upper right: Lateral relaxing incisions and nasal mucosa closure using the anterior triangular flap and lateral nasal mucosa flaps. Release of the abnormal muscular insertion is performed. But two flap palatoplasty can lengthen the soft palate by push-back
  Arms: group B

SUMMARY:
Cleft palate is one of the most common congenital abnormalities of the orofacial region throughout the world. This condition can cause facial deformity, feeding problems, frequent middle ear infections, dental defects, speech abnormalities and emotional problems . Early surgical repair of this congenital anomaly prevents the psychological and functional problems associated with the deformity . Patients may develop various complications after primary palatoplasty including palatal fistula and velopharyngeal insufficiency (VPI) which are relatively common .

The main goal of cleft palate repair is to achieve normal speech and adequate velopharyngeal function with minimal effect on facial growth. The primary objective in the surgical repair of a cleft palate is the development of normal speech. Speech quality remains the most important standard for assessing clinical outcomes and the success of surgical procedures. Many surgical techniques for palate correction have been described determining the most effective technique for the surgical repair of palatal clefts continues to cause controversy .

The incidence of VPI post cleft palate repair is 20-30% of patients . If there is significant velopharyngeal dysfunction during normal speech development, many children learn to compensate for the lack of intraoral pressure. They produce a hoarse voice because of vocal fold adduction and sudden release. Compared with the adductor vocal fold palsy .

ELIGIBILITY:
Inclusion Criteria:

* •children more than 3 years old

  * Type of cleft: isolated cleft palate

Exclusion Criteri

* Complicated cases by fistula or redo,
* Missed follow up; less than 6 months.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Velopharyngeal Insufficiency Evaluation | 20 months
  Velopharyngeal gap size in centimeters using nasopharyngoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wong FK, Hagg U. An update on the aetiology of orofacial clefts. Hong Kong Med J. 2004 Oct;10(5):331-6. PMID 15479962
- [Background] Donkor P, Bankas DO, Agbenorku P, Plange-Rhule G, Ansah SK. Cleft lip and palate surgery in Kumasi, Ghana: 2001-2005. J Craniofac Surg. 2007 Nov;18(6):1376-9. doi: 10.1097/01.scs.0000246504.09593.e4. PMID 17993884
- [Background] Abdaly H, Omranyfard M, Ardekany MR, Babaei K. Buccinator flap as a method for palatal fistula and VPI management. Adv Biomed Res. 2015 Jul 27;4:135. doi: 10.4103/2277-9175.161529. eCollection 2015. PMID 26322283
- [Background] Bishop A, Hong P, Bezuhly M. Autologous fat grafting for the treatment of velopharyngeal insufficiency: state of the art. J Plast Reconstr Aesthet Surg. 2014 Jan;67(1):1-8. doi: 10.1016/j.bjps.2013.09.021. Epub 2013 Sep 20. PMID 24090720